CLINICAL TRIAL: NCT06071130
Title: Emotion, Aging, and Decision Making
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePaul University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-2021-520
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Motivation; Aging; Health Behavior; Emotions; Social Behavior
MeSH Terms: conditions — Health Behavior; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experiment 4A & 4B (Experimental): Participants will attend for 3 sessions/week for 8 weeks. Instructors will conduct classes and maintain participant attendance records. Exercise components include flexibility, aerobics, strengthening, and physical activity logs. Classes begin and end with 10-minute warmups and cool downs. Participants are taught low-impact aerobic routines to maximize self-efficacy for physical activity maintenance after the program. This will include fitness walking that will progress from each participant's maximum capacity to the goal of 20 minutes of sustained walking. Participants will be instructed on how to gauge their exercise intensity and physical exertion. The strengthening focus of the program will improve independent functioning by targeting lower extremity strength with a graded, task-specific approach. Resistance will be progressively increased over the course of the program by adding weight. At the end of each exercise session, participants will log physical activity.
  Interventions: Behavioral: Fit and Strong

INTERVENTIONS:
Behavioral: Fit and Strong — Procedure: During Years 3-5, participants will be recruited in waves through our standard recruitment practices to participate in Experiments 4A at the City of Chicago park sites. We will first prescreen them via telephone to verify that potential participants meet the inclusion criteria. F&S! classes will be offered at two pre-determined Chicago park sites. Each of the two sites will host the 8-week-long program once in the spring and once in the fall for two years for a total of four F&S! cycles at each center (totaling 8 F&S! cohorts). Upon consenting to be in E4A, participants will be enrolled in F&S! at the site closest to their home or the wait-list control. In the pre-intervention phase, participants both in F&S! and on the waitlist will come to the lab at DePaul to complete the pre-intervention measurement batter. Within one week after baseline measurements, participants will attend F&S! for 3 sessions a week for 8 weeks.

SUMMARY:
Exercise is routinely recommended because of its benefits for physical, cognitive, and mental health. It is especially beneficial for older adults due to its potential buffering effects against Alzheimer's disease and related dementias (Luck et al., 2014). However, little is known about how to best encourage older adults to exercise. Based on behavior change theory, different intrapersonal and interpersonal motivational factors are likely to be relevant during the contemplation, action, and maintenance stages of behavior change. Generally, as a result of motivational shifts toward prioritizing positivity and socially meaningful goals with advancing age (Carstensen, 2006), socioemotional aspects of decision making may become more salient and influential for older adults (Mikels et al., 2015; Peter et al., 2011). Our previous work has demonstrated that positive affect (Mikels et al., 2020) and social goals (Steltenpohl et al., 2019) play a critical role in older adults' motivation to exercise, but these two lines of research have not been integrated to date. Recent work indicates that positive affect is particularly beneficial for health when shared in social connections (Fredrickson, 2016; Major et al., 2018), and the proposed work will, for the first time, examine how shared interpersonal positivity may impact exercise decision making and behavior, especially during the contemplation and action/maintenance stages of behavior change.

But who are the older adults that benefit the most from exercise in terms of physical, cognitive, and mental health (and should be hence be targeted with messages)? Not all older adults reap the benefits of exercise (Sparks, 2014) and, conversely, sedentary older adults have the most to gain. Overall, the current proposed research program is innovative in its (a) translational application of insights from affective, cognitive, and aging theory and research to understand the antecedents and outcomes of exercise decision making in younger and older adults, (b) conceptualization of both the social and emotional aspects of decision making, (c) development of novel methods for health messaging that incorporate social influences, and (d) novel assessments of the exercise-health link.

DETAILED DESCRIPTION:
Our specific aims are:

Aim 1: To understand how social and emotional processes contribute to age differences in health-related decision making. Message framing is an effective means of promoting behavior change, with loss-framing emphasizing the negative consequences of not engaging in a behavior, and gain-framing emphasizing the benefits of engaging in a behavior (Rothman & Salovey, 1997). Although affect has been examined in messaging, intrapersonal vs. interpersonal benefits and consequences as well as the role of shared positive affect have not. We propose that interpersonal vs. intrapersonal framing will differentially influence positivity toward exercise for sedentary and active older vs. younger adults. Experiment 1 (laboratory-based) will examine affective reactions, evaluations, and behavioral intentions in response to framed messages. To better understand the social processes involved in exercise decisions, Experiment 2 (field-based) will examine the same outcomes of Experiment 1 when people exercise alone or with another person, with a focus on whether shared positive affect is more motivating for older vs. younger adults when engaged in physical activity.

Aim 2: To determine how social and emotional factors impact exercise engagement, adherence, and maintenance. Experiments 3, 4A, and 4B will examine whether intrapersonal vs. interpersonal factors disproportionately impact exercise intentions and behavior. In Experiment 3, intrapersonal vs. interpersonal framing will be applied to recruit and enroll younger and older adults into an exercise program. In Experiment 4A, we will examine whether social and emotional factors - including shared positive affect - influence the engagement and adherence of older adults enrolled in an evidence-based fitness program, Fit & Strong! (Hughes et al., 2006). In Experiment 4B, we will measure social and emotional influences on continued physical activity one year after the program ends. In these latter two experiments, we will measure actual behavioral outcomes including objective measures of physical activity and attendance, as well as shared positive affect, cognitive function, and well-being.

Aim 3: To extend the established benefits of Fit & Strong! for older adults into physiological and cognitive domains. It is well-established that exercise improves physical, mental, and cognitive health (Hillman et al., 2008; Hughes et al., 2006). We will expand the documented benefits of a particular exercise intervention tailored for older adults, Fit & Strong!, by examining its impact on cardiovascular, somatic physiological, social, and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Experiment 4A: We will follow the standard exclusion protocol used in previous Fit & Strong! studies (e.g., Hughes et al., 2004; 2006). The participant's physician will be contacted for clearance to participate if they have a history of high blood pressure, or experience dizziness, lightheadedness, or chest pain or pressure during physical activities (walking, climbing stairs, and household chores, etc.) (see document: "E4_NeedforPhysicianScreeningQuestionnaire.docx"). Additionally, physicians will be contacted if participants indicate that they fall, feel unsteady, or use an assistive walking or standing device. For these conditions and any special considerations that a participant may express, physicians will be contacted for clearance.

Experiment 4B: Only participants who participated in Experiment 4A are eligible to participate in Experiment 4B.

Exclusion Criteria:

* Experiment 4A: We will follow the standard exclusion protocol used in previous Fit & Strong! studies (e.g., Hughes et al., 2004; 2006). For instance, participants will be excluded for joint steroid injections within 3 months, knee or hip surgery within the previous 6 months or next year, rheumatoid arthritis or other systemic inflammatory arthritis, or uncontrolled diabetes. The participant's physician will be contacted for clearance to participate if they have a history of high blood pressure, or experience dizziness, lightheadedness, or chest pain or pressure during physical activities (walking, climbing stairs, and household chores, etc.) (see document: "E4_NeedforPhysicianScreeningQuestionnaire.docx"). Additionally, physicians will be contacted if participants indicate that they fall, feel unsteady, or use an assistive walking or standing device. For these conditions and any special considerations that a participant may express, physicians will be contacted for clearance (see document: "StatementofMedicalClearanceforExercise.docx" and "CoverLetterforMedicalClearanceforExercise.docx").

Experiment 4B: Participants who did not participate in Experiment 4A are not eligible to participate in Experiment 4B.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-03 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Connecting Socioemotional Aspects of Exercise to Improvements in Physical Health among Older Adults | two years
  Materials & Measures for Pre- and Post-Intervention: The measurement battery will include: a basic demographic form, a cognitive battery in addition to several oral inductive reasoning measures: Letter Sets and Figure Classification, and Everyday Problem Solving. We will also administer measures of physical activity related variables that have been collected in previous Fit & Strong! studies, which include: a paper measure of self-efficacy for arthritis self-management, a paper measure of exercise adherence self-efficacy, an oral functional lower extremity muscle strength, 6-minute distance walk in which we measure how far a participant walks in 6 minutes, and a paper version of the Western Ontario and McMasters University Osteoarthritis Index.

CONTACTS AND LOCATIONS:
Locations (1):
- DePaul University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No